CLINICAL TRIAL: NCT02346214
Title: Smartphone Ophthalmoscope Lens Vascularity Estimated Gestational Age (SOLVE-GA)
Brief Title: Smartphone Ophthalmoscope of Lens Vascularity to Estimate Gestational Age
Status: Completed | Type: Observational
Sponsor: RTI International (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); Duke University (Other); Loma Linda University (Other); University of Iowa (Other)
Responsible Party: Sponsor
Other Study IDs: OPP1119360
Record Dates: First submitted 2015-01-20; First posted 2015-01-26 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Gestational Age
Keywords: Gestational Age; Anterior Lens Capsule Vascularity; Preterm; Method-comparison
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Preterm and term neonates: A. Preterm and term neonates B. Singleton live births between 26 and 42 weeks gestation (determined by first of early-second trimester ultrasound dating) at three referral hospitals

SUMMARY:
The purpose of this study is to develop a novel, highly automated method of gestational age estimation at delivery combining anterior lens capsule vascularity (ALCV) and biophysical parameters appropriate for use in low income countries. The specific aims of the proposed study are: (1) To develop an algorithm to predict gestational age at delivery from 26 to 42 weeks' gestation with ALCV and key biophysical parameters (2)To evaluate the performance of ALCV and biophysical parameter-based gestational age estimates. Specifically, we hypothesize that the accuracy of the predictive algorithm will be comparable to commonly used measures of gestational age dating (±2 days) and have better precision (±14 days) than commonly used measures of gestational age dating.

DETAILED DESCRIPTION:
Postnatal gestational age dating methods are needed in low/middle income settings as ultrasound is often unavailable, last menstrual dates uncertain, and physical/neurological scoring complex. The disappearance of anterior lens capsule vascularity (ALCV), a normal embryological process, has a high correlation with gestational age at delivery among preterm neonates. We will use an observational method-comparison study to establish the validity of smartphone ophthalmoscope ALCV gestational age estimates among preterm infants at delivery compared to the referent standard of ultrasound gestational age estimates. Study objectives and methods include the following: Objective 1. Develop an ALCV biomarker dataset from smartphone ophthalmoscope images using automated image analysis software. The dataset will include image features including: vessel quantity, lens clearing, tortuosity, vessel thickness, and branching angles and coefficients. Methods: (1) capture ALCV images via smartphone ophthalmoscope within 24 hours of delivery, and (2) segment ALCV images using software developed for the assessment of retinal vasculature. Proposed software will convert images into graphs and automatically find the vasculature based on the Dijkstra's shortest-path algorithm. The proposed software is tested for video-indirect neonatal ophthalmoscope images. Objective 2. Develop an algorithm to predict gestational age at delivery from 26 to 42 weeks' gestation with the ALCV biomarker dataset combined with key neonatal biophysical measures. Methods: (1) conduct descriptive and univariate analyses of predictors and assess linear model assumptions, and (2) fit a constrained linear regression model by selecting and shrinking estimated model coefficients from a fully specified model in the original sample to optimize predictive accuracy and model parsimony. Objective 3. Assess the performance of ALCV gestational age estimates compared to referent standard ultrasound estimates. Methods: (1) compare distributions of gestational age and the mean difference in days between dating methods, (2) test agreement between dating methods using Lin's concordance correlation coefficient and Bland-Altman plots with limits of agreement (3) internally validate test agreement using a bootstrap procedure for optimism correction of the agreement statistics. All statistical analyses will be performed in SAS 9.4 (SAS, Cary, North Carolina, USA).

ELIGIBILITY:
Inclusion Criteria:

* Gestational age 260/7 to 426/7 weeks (based on antenatal ultrasound <20 weeks gestation)

  * Chronological age <24 hours
  * Consent of the patient's parents or legal guardians

Exclusion Criteria:

* Fused eyelids
* Corneal opacity or cataract
* Obstetrical ultrasound performed at <20 weeks' gestation not performed/not available
* Known genetic/congenital anomalies
* Known coagulopathies
* Patients who, in the opinion of the attending physician or clinical study staff, are too medically unstable to participate in the study safely

Max Age: 24 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Singleton live births between 26 and 42 weeks' gestation (determined by first or early-second trimester ultrasound dating)
Sampling Method: Non-Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Anterior lens capsule vascularity estimated gestational age | Within 24 hours of delivery
  The gestational age is estimated by eye lens vascularity measurement

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Griffin, Ph.D. M.P.H., Principal Investigator — RTI International
Locations (3):
- United States (3):
  - Loma Linda University Children's Hospital, Loma Linda, California
  - University of Iowa Children's Hospital, Iowa City, Iowa
  - University of North Carolina at Chapel Hill North Carolina Children's Hospital, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Altman, D. G. and J. M. Bland (1983).
- [Background] Bland, J. M. and D. G. Altman (2010).
- [Background] Blencowe, H., S. Cousens, D. Chou, M. Oestergaard, L. Say, A.-B. Moller, M. Kinney and J. Lawn (2013).
- [Background] Concato, J., P. Peduzzi, T. R. Holford and A. R. Feinstein (1995). Estrada, R., C. Tomasi, M. T. Cabrera, D. K. Wallace, S. F. Freedman and S. Farsiu (2011).
- [Background] Estrada, R., C. Tomasi, M. T. Cabrera, D. K. Wallace, S. F. Freedman and S. Farsiu (2012).
- [Background] Hittner HM, Gorman WA, Rudolph AJ. Examination of the anterior vascular capsule of the lens: II. Assessment of gestational age in infants small for gestational age. J Pediatr Ophthalmol Strabismus. 1981 Mar-Apr;18(2):52-4. doi: 10.3928/0191-3913-19810301-12. PMID 7195426
- [Background] Hittner HM, Hirsch NJ, Rudolph AJ. Assessment of gestational age by examination of the anterior vascular capsule of the lens. J Pediatr. 1977 Sep;91(3):455-8. doi: 10.1016/s0022-3476(77)81324-3. PMID 894419
- [Background] Nagpal J, Kumar A, Ramji S. Anterior lens capsule vascularity in evaluating gestation in small for gestation neonates. Indian Pediatr. 2004 Aug;41(8):817-21. PMID 15347869